CLINICAL TRIAL: NCT05186064
Title: Glioblastoma Targeted Treatment Option Maximization by Whole Genome Sequencing
Brief Title: Glioblastoma Targeted Treatment Option Maximization by WGS
Acronym: GLOW
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: UMC Utrecht (Other)
Collaborators: Amsterdam University Medical Center (Other); The Netherlands Cancer Institute (Other); The Elisabeth-TweeSteden Hospital (Other); Erasmus Medical Center (Other); Medical Center Haaglanden (Other); Isala (Other); Leiden University Medical Center (Other); Maastricht University Medical Center (Other); Medisch Spectrum Twente (Other); Radboud University Medical Center (Other); University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Dr. F.Y.F.L. de Vos, medical oncologist, UMC Utrecht
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NL79220.058.21 / N21.115
Record Dates: First submitted 2021-12-23; First posted 2022-01-11 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Glioblastoma
Keywords: first recurrence; whole genome sequencing
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- whole genome sequencing after standard of care resection at first relapse (Experimental)
  Interventions: Diagnostic Test: whole genome sequencing

INTERVENTIONS:
Diagnostic Test: whole genome sequencing — whole genome sequencing will be performed on tumor material after re-resection per standard of care

SUMMARY:
In Dutch centers performing neurosurgery on and/or treating GBM, all recurrent GBM patients are discussed in local tumor boards and this setup will be used to effectively identify possible GLOW study candidates. 160 patients that will undergo re-resection in the GLOW study will be presented with WGS results leading to added treatment options.

DETAILED DESCRIPTION:
Rationale: Glioblastoma (GBM), the most common primary brain tumor, is without exception lethal. Every year 1000 patients are diagnosed with this disease in the Netherlands. Despite neurosurgery, chemo -and radiation therapy, these tumors inevitably recur. Currently, there is no gold standard at time of recurrence and treatment options are limited. In a retrospective study in two Dutch neuro-oncology centers, the overall survival (OS) for patients with recurrent GBM receiving best supportive care was 3 months, while patients receiving systemic treatment (usually nitrosurea), radiation therapy or surgery followed by systemic treatment or radiotherapy had respectively 7.3 months, 9.2 months and 11 months OS. Unfortunately, the results of dedicated trials with new drugs have been very disappointing. For those to be meaningful, extensive molecular screening is needed.

The goal of the project is to obtain the evidence for changing standard of care procedures to include extensive molecular diagnostics and consequently adapt care guidelines for this specific patient group with very poor prognosis by offering optimal and timely benefit from novel therapies, even in the absence of traditional registration trials for this small volume cancer indication.

Objective: To determine the value of and generate the clinical evidence for routine application of Whole Genome Sequencing (WGS)-based diagnostics and targeted therapy guidance for glioblastoma patients at time of first recurrence.

Study design: Prospective diagnostic multicenter cohort study Study population: Adult glioblastoma patients with recurrent disease that are undergoing resection or debulking as part of their standard care and from whom written informed consent is obtained.

Intervention: A 10 mL blood sample will be drawn once to assess each patient's germline DNA background variation that will discriminate somatic mutations from the patient's germline DNA background variations. All other interventional procedures required to perform this study are part of standard procedures.

Main study parameters/endpoints:

Primary study endpoint: Overall survival

Secondary study endpoints:

* Tumor and blood collection success rate (target >85% of all patients included)
* Number of successful WGS reports (reports for >80% of patients for which tumor material was collected)
* Number of targeted treatment options identified (at least one potentially actionable DNA alteration in >75% of patients with a WGS report)
* Number of experimental treatments available for GBM patients (relevant (off-label) drugs for at least 50% of the identified indications should be available through a study, including the Drug Rediscovery Protocol (DRUP)
* Thirty-two percent of patients starting a targeted treatment in presence of actionable variant (currently 16%)

ELIGIBILITY:
Inclusion Criteria:

1. Histopathologically confirmed IDH wild type glioblastoma, first recurrence after standard chemoradiation; suitable for standard-of-care re-resection;
2. Age ≥ 18 years;
3. Able and willing to give written informed consent;
4. Life expectancy >3 months, allowing adequate follow-up of toxicity evaluation and antitumor activity;
5. KPS performance status ≥70.

Exclusion Criteria:

1. Currently actively treated in another antitumor clinical trial (excluding DRUP and STELLAR studies);
2. Patients with any other clinically significant medical condition which, in the opinion of the treating physician, makes it undesirable for the patient to participate in medication studies or which could jeopardize compliance with study requirements including, but not limited to ongoing or active infection, significant uncontrolled hypertension, or severe psychiatric illness/social situations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2022-07-25 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
overall survival | 3 years

SECONDARY OUTCOMES:
number targeted treatment options identified | 2 years
percent of patients starting a targeted treatment in presence of actionable variant | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Haaglanden Medisch Centrum, The Hague, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] van Opijnen MP, Broekman MLD, de Vos FYF, Cuppen E, van der Hoeven JJM, van Linde ME, Compter A, Beerepoot LV, van den Bent MJ, Vos MJ, Fiebrich HB, Koekkoek JAF, Hoeben A, Kho KH, Driessen CML, Jeltema HR, Robe PAJT, Maas SLN. Study protocol of the GLOW study: maximising treatment options for recurrent glioblastoma patients by whole genome sequencing-based diagnostics-a prospective multicenter cohort study. BMC Med Genomics. 2022 Nov 4;15(1):233. doi: 10.1186/s12920-022-01343-4. PMID 36333718